CLINICAL TRIAL: NCT00203918
Title: Prostate Cancer Utilities and Cost-Effectiveness Analysis
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 12843B
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Cost-Effectiveness Analysis; Utility Assessment
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prostate biopsies: Males undergoing prostate biopsies
  Interventions: Behavioral: Survey, interview; Behavioral: patient utility scores (i.e. patient preference weights)

INTERVENTIONS:
Behavioral: Survey, interview — A survey is administered to patients visiting the urology clinic to undergo prostate biopsies to validate a method of utility assessment, and understand patients' individual evaluations of treatment-related health states. Medical records will also be reviewed 00 days after the survey was administered to determine whether this data reflects actual treatment decisions.
Behavioral: patient utility scores (i.e. patient preference weights) — comparison of patient preferences

SUMMARY:
The purpose of this study is to help doctors and patients make better decisions about prostate cancer treatment. This research is being done because we do not know how patient preferences for health states related to prostate cancer affect the final treatment decision.

DETAILED DESCRIPTION:
The goal of this project is to incorporate patients' preferences into a previously developed prostate cancer treatment decision-model and to understand the implications for doing so for cost-effectiveness analysis. To do this, it is first necessary to obtain patient utility scores (i.e., patient preference weights). To do this we will perform a survey of patients visiting the urology clinic to undergo prostate biopsies to validate a method of utility assessment, and understand the patients' individual evaluations of treatment-related health studies. We will also ask patients questions relating to their anxiety levels concerning the possible diagnosis of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing prostate biopsy

Exclusion Criteria:

* Women and children will be excluded, as prostate cancer occurs in men only
* Diagnosis of dementia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients visiting the urology clinic at the University of Chicago.
Sampling Method: Probability Sample
Enrollment: 481 (Actual)
Dates: Start 2004-01; Primary Completion 2011-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Utility scores for treatment outcomes | 90 days after enrollment
  Patient utility scores (i.e. patient preference weights) are calculated using survery data will determine which prostate cancer treatment would be most cost-effective for each subject. Patients will be contacted by phone and patient records will be reviewed 90 days after the survey has been completed to determine whether this data reflects actual treatment decisions.

SECONDARY OUTCOMES:
Anxiety levels | 90 days after enrollment
  We will also ask patients questions relating to their anxiety levels concerning the possible diagnosis of prostate cancer.

CONTACTS AND LOCATIONS:
Overall Officials: David Meltzer, M.D., Ph.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States